CLINICAL TRIAL: NCT06593366
Title: A Pilot Feasibility Randomized Controlled Trial of Fecal Microbiota Transplant for Adolescent Anorexia Nervosa
Brief Title: Fecal Microbiota Transplant for Anorexia Nervosa
Acronym: FMT-AN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Jennifer Couturier, Associate Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: FMTAN
Record Dates: First submitted 2024-07-26; First posted 2024-09-19 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Anorexia Nervosa Restricting Type; Anorexia Nervosa; Anorexia in Adolescence; Anorexia in Children; Anorexia
Keywords: anorexia nervosa; fecal microbiota transplant; pilot study; randomized controlled trial; feasibility
MeSH Terms: conditions — Anorexia Nervosa; Anorexia | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties will be blinded to the participant's treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecal Microbiota Transplant (Active Comparator): Banked donor stools that have been previously screened, prepared and frozen per previous protocols will be used to prepare all oral FMT capsules (OFC) through the laboratory of a collaborator. Recipients will receive OFC (two capsules, twice a day, twice per week) prepared from a single donor throughout their 8-week treatment course, to support assessment of FMT engraftment in recipients; this totals to 64 capsules across the duration of the study. Each OFC will contain approximately 15.0g of dried healthy donor stool contained within a size 00 gelatin capsule.
  Interventions: Biological: Fecal Microbiota Transplant
- Placebo (Placebo Comparator): Matching oral placebo capsules (OPC) containing methylcellulose will be identical in terms of size, colour, taste, and dosing. Participants will be asked to take the Placebo treatment capsules twice a day for two days per week for a duration of eight weeks (total 64 capsules).
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Fecal Microbiota Transplant — An investigational biologic comprised of 15.0g of dried healthy donor stool contained within a size 00 gelatin capsule, to be taken twice per day, twice per week over an 8-week duration.
  Arms: Fecal Microbiota Transplant
Drug: Placebo — Oral placebo capsules (OPC) containing methylcellulose, to be taken twice per day, twice per week over an 8-week duration.
  Arms: Placebo

SUMMARY:
The purpose of this pilot randomized-controlled trial is to determine whether Fecal Microbiota Transplant (FMT) treatment demonstrates feasibility, acceptability, and prelinary effectiveness among patients with anorexia nervosa (AN). Specifically, the investigators aim to compare changes in weight, gut microbiome, urine, blood biomarkers and mood symptoms between participants receiving the FMT intervention and placebo.

DETAILED DESCRIPTION:
In the following pilot randomized-controlled trial, the investigators' aim is to determine whether FMT treatment demonstrates feasibility, acceptability, and preliminary effectiveness in pediatric AN participants. The investigators will assess how the use of FMT affects participants' rate of weight restoration, gut microbiome, relevant urine and blood biomarkers, and mood symptoms. The investigators' rationale for performing the study is to better understand the interactions between the intestinal microbiome, energy regulation, and behavior. This will be the first study to assess the role of FMT in pediatric AN and will help establish whether this adjunctive treatment modality has benefit in managing the metabolic and behavioral manifestations of this complex neuropsychiatric disorder.

In terms of study procedures, members of a pilot sample of 20 AN patients recruited from McMaster Children's Hospital will be randomized to receive FMT or placebo. All participants will be asked to complete a battery of assessments at regular intervals over the 8-week intervention period, and at a follow-up point at four weeks post-intervention.

The study's primary outcomes are recruitment and retention rates. Descriptive statistics will be used to determine the number of adolescents who will agree to participate in the study and those who will complete the study.

One of the study's secondary outcomes is participants' attitudes toward FMT. This will be measured through qualitative interviews among those who completed the intervention and those who do not agree to participate in the study.

The investigators will know we have reached saturation by using a method called "information power" and will explore how broad the research questions are, if there are clear theories to guide the analysis, how varied the participants in the study are, and how much useful information is accrued. Based on this, the investigators will determine the appropriate number of interviews to lead.

The remaining secondary outcome is a battery of preliminary outcomes (clinical, biological, biochemical and safety). The investigators will assess these outcomes at multiple timepoints using questionnaires, anthropometric data, stool analysis (16s rRNA), urine metabolic analysis, saliva ultra filtrates, changes in blood work, and common terminology criteria for adverse events for safety outcomes.

ELIGIBILITY:
Inclusion Criteria: All study subjects will have been diagnosed with AN (restricting type or binge eating/purging type) by the primary physician on the ED team, as per standard approach. Study participants will:

* Be 12-17 years-old at time of recruitment
* Have capacity to consent
* Be assigned female sex at birth (may be gender diverse)
* Be active patients in the pediatric ED program at MCH
* Have a weight that is <85% of the Treatment Goal Weight, as determined by the treating physician

Exclusion Criteria: Potential study subjects will be excluded due to the following reasons:

* Exposure to antibiotics within two weeks of study randomization
* Initiation of new probiotics / oral nutritional supplements within two weeks of randomization
* Active pregnancy
* Active psychosis or suicidal ideation
* Other comorbidities that may affect weight or the gut microbiome including celiac disease, inflammatory bowel disease (or other conditions as determined by the study team)

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Through study completion, an average of one year.
  The number of participants who are consented into the study divided by the number of participants who show interest in the study.
Retention Rate | Through study completion, an average of one year.
  The number of participants who completed the study divided by the number of participants consented into the study.

SECONDARY OUTCOMES:
Attitudes towards Fecal Microbiota Transplant | Week 12 (follow-up)
  Attitudes towards FMT will be studied via semi-structured qualitative interviews of all participants: the 20 adolescents and their parents in the trial, and the 10 adolescents and their parents who decline participation, and their guardians. Using Qualitative Description, interviews will explore patient and guardian attitudes toward FMT, as well as their impressions of efficacy (if they participated in the trial). Questions will include perceptions of "natural" versus "drug" products, perspectives on causes of AN, and interests in other potential treatments. Interviews will be conducted virtually, using Zoom for Healthcare, transcribed verbatim and then coded for themes using NVivo. This analysis stays close to the data with little to no interpretation. Our analysis will also include a summative content analysis.
Height | Week 0 (baseline), Week 4 (mid-treatment), Week 8 (post-intervention), Week 12 (follow-up)
  Height will be collected.
Weight | Week 0 (baseline), Week 2, Week 4 (mid-treatment), Week 6, Week 8 (post-intervention), Week 10, Week 12 (follow-up)
  Weight will be measured between hospital visits using home weight scales provided to study participants.
Eating Disorder Examination Questionnaire | Week 0 (baseline), Week 4 (mid-treatment), Week 8 (post-intervention), Week 12 (follow-up)
  The EDEQ is a 28-item standardized questionnaire that measures the severity of symptoms of eating disorders, including menstrual status.
Beck Depression Inventory | Week 0 (baseline), Week 4 (mid-treatment), Week 8 (post-intervention), Week 12 (follow-up)
  The BDI is a 21-item questionnaire used to measure the severity of depressive symptoms.
Beck Anxiety Inventory | Week 0 (baseline), Week 4 (mid-treatment), Week 8 (post-intervention), Week 12 (follow-up)
  The BAI is a 21-item questionnaire used to measure the severity of anxiety symptoms.
Yale-Brown-Cornell Eating Disorder Scale | Week 0 (baseline), Week 4 (mid-treatment), Week 8 (post-intervention), Week 12 (follow-up)
  The YBC-EDS assesses impairment, persistence and degree of obsessional thinking and compulsiveness about eating behaviors.
Gastrointestinal Symptom Rating Scale | Week 0 (baseline), Week 4 (mid-treatment), Week 8 (post-intervention), Week 12 (follow-up)
  This is a 15-item rating scale to capture a variety of GI symptoms.
Changes in stool metabolites | Week 0 (baseline), Week 4 (mid-treatment), Week 8 (post-intervention), Week 12 (follow-up)
  Stool will be collected in to examine changes in alpha- and beta- diversity of microbiota, as well as engraftment of donor specific strains/genes and microbially-derived metabolite levels throughout the study. All stool samples will be collected using an at-home collection kit. Samples will be collected and stored in locked, secure -80°C study freezers upon being brought to the hospital or shipped by paid courier by participants. Stool samples will be sequenced for 16s rRNA gene profiling. All 16s rRNA analyses will be performed using in-house bioinformatics pipelines through the laboratory of a collaborator to identify amplicon sequence variants, perform taxonomic assignments, and analyze alpha- and beta-diversity and differential taxonomic abundance.
Changes in urine metabolomics | Week 0 (baseline), Week 4 (mid-treatment), Week 8 (post-intervention), Week 12 (follow-up)
  Urine samples will be collected from each participant. Nontargeted metabolite profiling is a method used to explore and identify as many metabolites as possible in a sample to identify whatever is present. This approach is designed to help discover new metabolites, and identify changes in metabolite levels that may correlate with other outcomes. We will report differences in highest-abundance metabolites using t-tests to compare their presence between groups, and correlation coefficients to identify associations between outcomes.
Changes in saliva ultrafiltrates | Week 0 (baseline), Week 4 (mid-treatment), Week 8 (post-intervention), Week 12 (follow-up)
  Saliva samples will be collected for metabolomic analysis. Saliva ultrafiltrates will be analyzed as described above for stool and urine samples by a collaborator. All saliva ultrafiltrates will be reported using the same multisegment injection-capillary electrophoresis-mass spectrometer, where metabolites are reported using effect sizes to compare relative concentrations against reference standards.
Changes in complete blood count | Week 0 (baseline), Week 8 (post-intervention)
  Using the provided blood samples, changes in complete blood count from baseline to post-intervention will be compared using paired t-tests. The complete blood count includes (with their measurement units):
  Red blood count (RBC)- cells/L Hemoglobin (Hb)- g/L Hematocrit- L/L Mean corpuscular volume (MCV)- fL Mean Corpuscular Hemoglobin (MCH)- pg Mean corpuscular hemoglobin concentration (MCHC)- g/L Red cell distribution width (RDW)- % White blood count (WBC) - cells/L Neutrophils - cells/L Lymphocytes - cells/L Eosinophils - cells/L Basophils - cells/L Monocytes - cells/L
Changes in C-reactive protein | Week 0 (baseline), Week 8 (post-intervention)
  Using the provided blood samples, changes in C-reactive protein (CRP) from baseline to post-intervention will be compared using paired t-tests. CRP (measured in mg/L) is used to monitor inflammation in acute or chronic conditions.
Changes in alkaline phosphatase | Week 0 (baseline), Week 8 (post-intervention)
  Using the provided blood samples, changes in alkaline phosphatase (ALP) from baseline to post-intervention will be compared using paired t-tests. ALP (measured in U/L) is associated with liver function.
Changes in alanine aminotransferase | Week 0 (baseline), Week 8 (post-intervention)
  Using the provided blood samples, changes in alanine aminotransferase (ALT) from baseline to post-intervention will be compared using paired t-tests. ALT (measured in U/L) is associated with liver function.
Changes in 25-OH Vitamin D | Week 0 (baseline), Week 8 (post-intervention)
  Using the provided blood samples, changes in 25-OH Vitamin D from baseline to post-intervention will be compared using paired t-tests. 25-OH Vitamin D (measured in ng/ml) is used as a measure of Vitamin D levels.
Changes in albumin | Week 0 (baseline), Week 8 (post-intervention)
  Using the provided blood samples, changes in albumin from baseline to post-intervention will be compared using paired t-tests. Albumin (measured in g/L) is associated with liver and kidney function.
Changes in follicle stimulating hormone | Week 0 (baseline), Week 8 (post-intervention)
  Using the provided blood samples, changes in follicle stimulating hormone (FSH) from baseline to post-intervention will be compared using paired t-tests. FSH (measured in mIU/mL) is important for determining aspects of fertility and menstruation.
Changes in luteinizing hormone | Week 0 (baseline), Week 8 (post-intervention)
  Using the provided blood samples, changes in luteinizing hormone (LH) from baseline to post-intervention will be compared using paired t-tests. LH (measured in IU/L) is important for determining aspects of fertility and menstruation.
Changes in free testosterone | Week 0 (baseline), Week 8 (post-intervention)
  Using the provided blood samples, changes in free testosterone from baseline to post-intervention will be compared using paired t-tests. Free testosterone (measured in nmol/L) is important for assessing various bodily functions related to hormones.
Presence of safety outcomes | Through study completion, an average of one year.
  Common Terminology Criteria for Adverse Events (CTCAE) will be used to define adverse events and serious adverse events. This framework will be used to classify broad safety concerns throughout our trial.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Couturier, MD, MSc, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data to other researchers.